CLINICAL TRIAL: NCT05447559
Title: Multicentre, Adaptive, Double-blind, Three-arm, Placebo-controlled, Noninferiority Trial Examining Antimicrobial Prophylaxis Duration in Cardiac Surgery
Brief Title: Duration of Cardiac Antimicrobial Prophylaxis Outcomes Study
Acronym: CALIPSO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: The Australian and New Zealand College of Anaesthetists (ANZCA) (Unknown)
Responsible Party: Principal Investigator, Trisha Nicole Peel, Professor Trisha Peel, Monash University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 228/22
Record Dates: First submitted 2022-06-27; First posted 2022-07-07 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Surgical Site Infection
Keywords: Cardiac surgery
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cefazolin; Water; Injections

STUDY DESIGN:
Intervention Model Description: Adaptive, double-blind, three-arm, placebo-controlled, phase IV, noninferiority trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, treating clinicians, all members of the research team including the study statistician will be blinded to treatment arm allocation.
  Active treatment will consist of 2-grams cefazolin powder for injection. Placebo will consist of an identical empty vial. The commercial labels will be removed and a sheath placed over the vial. Amber-tinted syringes will be provided for drawing up and administration of cefazolin/placebo to mask study arm.
  The vial containing cefazolin or placebo will be reconstituted in a minimum of 10 mL of sterile water for injections and administered in keeping with product information for cefazolin and / or local guidelines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intraoperative only Surgical Antimicrobial Prophylaxis Arm (Placebo Comparator): Placebo administered every 8-hours following the preoperative dose (time=0) for a total of five postoperative doses
  Interventions: Drug: Water for injection
- Intraoperative and 24-hours Postoperative Surgical Antimicrobial Prophylaxis Arm (Other): Cefazolin (2g) administered 8-hourly following the preoperative dose (time=0) for two doses then placebo 8-hourly for three doses (total of 5 postoperative doses of cefazolin/placebo)
  Interventions: Drug: Cefazolin; Drug: Water for injection
- Intraoperative and 48-hours Postoperative Surgical Antimicrobial Prophylaxis Arm (Active Comparator): Cefazolin (2g) administered every 8-hours following the preoperative dose (time=0) for a total of five postoperative doses
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Cefazolin — Intravenous administration of 2 g cefazolin
  Arms: Intraoperative and 24-hours Postoperative Surgical Antimicrobial Prophylaxis Arm; Intraoperative and 48-hours Postoperative Surgical Antimicrobial Prophylaxis Arm
Drug: Water for injection — Intravenous administration of 10mL sterile water for injection
  Arms: Intraoperative and 24-hours Postoperative Surgical Antimicrobial Prophylaxis Arm; Intraoperative only Surgical Antimicrobial Prophylaxis Arm

SUMMARY:
This multicentre, adaptive, pragmatic, double-blind, three-arm, placebo-controlled, randomised, non-inferiority clinical trial will compare the incidence of surgical site infection and other healthcare associated infections, health economic and microbiological impact after intraoperative only (Arm A), to 24 hours (Arm B) and, to 48 hours (Arm C) of IV cefazolin and placebo postoperative surgical antimicrobial prophylaxis in patients undergoing cardiac surgery

DETAILED DESCRIPTION:
This trial will evaluate the clinical effectiveness, health-economic outcomes and microbiological impact of intraoperative (only) compared with intraoperative plus postoperative prophylaxis durations in patients undergoing cardiac surgery.

CALIPSO, a multicentre, adaptive, double-blind, three-arm, placebo-controlled, phase IV, noninferiority trial will examine the incidence proportion of SSI following cardiac surgery. Our three-intervention trial will compare:

Arm A Administration of prophylaxis in intraoperative period only Arm B Administration of prophylaxis in intraoperative plus for 24 hours postoperatively Arm C Administration of prophylaxis in intraoperative plus for 48 hours postoperatively

ELIGIBILITY:
Inclusion Criteria:

- Adult patients undergoing cardiac surgery involving a median sternotomy

Exclusion Criteria:

* Age <18 years
* American Society of Anesthesiology (ASA) 5
* Subjects with GFR <40mL/min/1.73m2 or those requiring continuous renal replacement therapy, haemodialysis or peritoneal dialysis
* Surgery for suspected or proven endocarditis or deep sternal wound infection
* Documented cefazolin hypersensitivity
* Documented methicillin resistant Staphylococcus aureus (MRSA) colonisation or infection in the 12-months prior to index surgery
* Cardiac transplantation
* Procedures involving insertion ventricular assist device or mechanical circulatory support device
* Procedures not involving a median sternotomy
* Patients previously enrolled and randomised to the CALIPSO trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9180 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of surgical site infection | 90 days from index surgery
  Surgical site infection according to CDC / NHSN definition

SECONDARY OUTCOMES:
Incidence of Clostridioides difficile infection | 30 days from index surgery
  Clostridioides difficile infection according the CDC definitions
Incidence of other health care association infections | From date of randomization until the date of discharge from the acute healthcare facility or date of death from any cause, whichever came first, assessed up to 30 days from index surgery
  Composite of all other HCAIs (pneumonia, blood stream infection and urinary tract infection)

OTHER OUTCOMES:
Incidence of Antimicrobial hypersensitivity reactions | From date of randomization until the date of discharge from the acute healthcare facility or date of death from any cause, whichever came first, assessed up to 30 days from index surgery
  Immediate (<48 hrs after exposure) or delayed (≥24 hrs after exposure) reaction to study drug
All-cause mortality rate | 180 days from index surgery
  Death reported up to 180 days from index cardiac surgery due to any cause.
Incidence of acute kidney injury | From date of randomization until the date of discharge from the acute healthcare facility or date of death from any cause, whichever came first, assessed up to 30 days from index surgery
  AKI will be defined according to the RIFLE criteria
Incidence of surgical site infections due to drug-resistant infections | 90 days from index surgery
  Surgical site infections due to drug-resistant infections (defined as resistance to cefazolin)

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Peel, MBBS GradCertRes FRACP PhD, Principal Investigator — Monash University
Locations (22):
- Australia (19):
  - Westmead Hospital, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Adelaide, South Australia
  - Flinders Private, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria
  - Epworth HealthCare, Melbourne, Victoria
  - Epworth Eastern HealthCare, Melbourne, Victoria
  - Cabrini Health, Melbourne, Victoria
  - Victorian Heart Hospital, Melbourne, Victoria
  - Sir Charles Gairdner, Nedlands, Western Australia
  - St John of God Subiaco Hospital, Perth, Western Australia
  - Fiona Stanley Hospital, Perth, Western Australia
  - St Vincent's Hospital, Melbourne
- New Zealand (3):
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Wellington

IPD SHARING:
Plan to Share IPD: No